CLINICAL TRIAL: NCT06131996
Title: Comparison of the Effects of Volar-assisted and Elastic Wrist Splints on Edema, Pain, Grip Strength and Functionality in Pregnant Women With Carpal Tunnel Syndrome
Brief Title: The Effect of Splints in Pregnant Women With Carpal Tunnel Syndrome
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Mardin Artuklu University (Other)
Responsible Party: Principal Investigator, Funda Mete Cavus, Principal Investigator, Mardin Artuklu University
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: 2021/007
Record Dates: First submitted 2023-11-02; First posted 2023-11-15 (Actual); Last update posted 2023-11-15 (Actual); Status verified 2023-11

CONDITIONS: Carpal Tunnel Syndrome; Pregnancy Related; Splints
MeSH Terms: conditions — Carpal Tunnel Syndrome

STUDY DESIGN:
Who Masked: Outcomes Assessor
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Volar-assisted splint group (Active Comparator): Participants used volar supported splint during sleep for 4 weeks. Exercise was performed at home for a total of 12 sessions, three sessions per week.
  Interventions: Other: Volar supported splint
- Elastic splint group (Active Comparator): Participants used velastic splint during sleep for 4 weeks. Exercise was performed at home for a total of 12 sessions, three sessions per week.
  Interventions: Other: elastic splint

INTERVENTIONS:
Other: Volar supported splint — participants used volar supported splint during sleep for 4 weeks. Exercise was performed at home for a total of 12 sessions, three sessions per week.
  Arms: Volar-assisted splint group
Other: elastic splint — participants used velastic splint during sleep for 4 weeks. Exercise was performed at home for a total of 12 sessions, three sessions per week
  Arms: Elastic splint group

SUMMARY:
It is aimed to compare the effect of two different splints on carpal tunnel syndrome in pregnant individuals after 4 weeks of use.

DETAILED DESCRIPTION:
Carpal tunnel syndrome (CTS) is a common musculoskeletal problem in pregnancy. The aim of this study is to compare the effects of rigid and elastic wrist splints on edema, pain levels, grip strength, and upper extremity functionality in pregnant women with CTS.

Pregnant women in the last trimester of pregnancy who were diagnosed with CTS were included in the study.

ELIGIBILITY:
Inclusion Criteria:

* Being in the last trimester of pregnancy,
* Having a diagnosis of CTS,
* Positive Tinnel and Phalen tests,
* Pain, tenderness, and numbness symptoms in the median nerve neurodynamic test,
* pain of at least 4 severity according to VAS,
* Edema due to pregnancy

Exclusion Criteria:

* Individuals in the 1st or 2nd trimester of pregnancy,
* Those with pain complaints below 4 according to VAS,
* Those with a history of CTS before pregnancy,
* Those who had undergone surgery in the hand-wrist region
* Those diagnosed with cervical disc herniation

Min Age: 18 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Gender Based: Yes — Individuals who are pregnant
Enrollment: 41 (Actual)
Dates: Start 2022-02-01 (Actual); Primary Completion 2022-10-01 (Actual); Study Completion 2022-12-30 (Actual)

PRIMARY OUTCOMES:
Quick Disabilities of the Arm, Shoulder, and Hand (Q-DASH) | before intervention and 4 weeks after intervention
  Q-DASH questionnaire is applied to evaluate upper extremity-related functionality and symptoms. Each item provides 5 response options and the overall score is calculated from the item scores. 0, no loss of function; 100 is interpreted as the most severe loss of function.
The Boston Questionnaire (BA) | before intervention and 4 weeks after intervention
  The Boston Questionnaire (BA) is specific to Carpal Tunnel Syndrome (CTS) and consists of two different scales that evaluate symptom severity and functional capacity.The scoring of each item varies between 1 and 5. The average score is obtained by dividing the total score by the number of items and ranges from 1 to 5. A high score indicates low functional capacity. Mean scores are calculated separately for symptom severity and functional capacity. The symptom score consists of 11 items and the function score consists of 8 items.
Grip strength | before intervention and 4 weeks after intervention
  Grip strength was measured with the Jamar hand dynamometer, which is recommended by the American Association of Hand Therapists (AETD) and whose validity and reliability have been confirmed in many studies.According to the measurement procedure, three repeated measurements were made for hand grip strength and the results were recorded in kilograms.
Volumetric measurement | before intervention and 4 weeks after intervention
  The water flooding method, which is considered the gold standard in the measurement of extremity volume and is preferred in the evaluation of edematous hand or foot volume, was used in this study.With this measurement method, the amount of overflowing water volume between the affected and unaffected extremities was compared and the amount of edema was determined.
Visual Analog Scale (VAS) | before intervention and 4 weeks after intervention
  The pain levels were measured by the Visual Analog Scale (VAS).It is scored between 0-10 cm. A high score indicates high pain.

CONTACTS AND LOCATIONS:
Overall Officials: Funda CAVUS, Study Director — MARDİN ARTUKLU UNİVERSİTY, VOCATIONAL SCHOOL OF HEALTH SERVICES,
Locations (1):
- Mardin Artuklu University, Mardin, Turkey (Türkiye)

IPD SHARING:
Plan to Share IPD: No